CLINICAL TRIAL: NCT05778422
Title: Comparative Study Between Pulsed Radiofrequency in Suprascapular Nerve or Bupivacaine Block for Chronic Shoulder Pain
Brief Title: Bupivacaine or Radiofrequency for Shoulder Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Leonardo Henrique Cunha Ferraro, Professor, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Bupivacaine x RF for shoulder
Record Dates: First submitted 2023-01-27; First posted 2023-03-21 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Shoulder Pain; Rotator Cuff Impingement Syndrome; Impingement Syndrome; Adhesive Capsulitis; Rotator Cuff Injuries
Keywords: shoulder pain; Pulsed radiofrequency; Bipuvacaine; Nerve block
MeSH Terms: conditions — Shoulder Pain; Shoulder Impingement Syndrome; Bursitis; Rotator Cuff Injuries | interventions — Anesthetics, Local; Pulsed Radiofrequency Treatment

STUDY DESIGN:
Intervention Model Description: Group 1 - pulsed radiofrequency Group 2 - bupivacaine
Who Masked: Outcomes Assessor
Masking Description: Participants were allocated to groups using a random sequence of numbers generated by computer using the Randomizer® program (www.random.org). The number of patients and the groups to which they would belong were randomly drawn. These numbers were placed in envelopes numbered from 1 to 40, which were drawn on the day of the consultation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pulsed Radiofrequency (Active Comparator): The investigators performed pulsed radiofrequency in the suprascapular nerve
  Interventions: Procedure: Pulsed radiofrequency
- Bupivacaine (Active Comparator): The investigators performed a blocade with bupivacaine in the suprascapular nerve.
  Interventions: Drug: Suprascapular nerve block with bipuvacaine

INTERVENTIONS:
Drug: Suprascapular nerve block with bipuvacaine — Suprascapular nerve block with Bipuvacaine: a 50mm 22G needle (Stimuplex, BBraun) was introduced up to the suprascapular fossa, guided by ultrasound, and the location was confirmed by motor stimulation with contraction of the supraspinatus and infraspinatus muscles. Next, 5 ml of 0.25% bupivacaine with adrenaline was injected.
  Other Names: Suprascapular nerve block with local anesthetic
  Arms: Bupivacaine
Procedure: Pulsed radiofrequency — After confirming the location, the needle mandrel was removed and the radiofrequency cannula was introduced through the needle, 2ml of 1% lidocaine without epinephrine was injected, followed by application of pulsed radiofrequency for 180sec at 42°C by radiofrequency (radiofrequency generator system BMS-50N, Bramsys).
  Other Names: Pulsed radiofrequency in suprascapular nerve
  Arms: Pulsed Radiofrequency

SUMMARY:
Comparative study between pulsed radiofrequency in suprascapular nerve or bupivacaine block for chronic shoulder pain

DETAILED DESCRIPTION:
Prospective, randomized, comparative study of 40 participants with chronic shoulder pain allocated into two groups. Patients in group 1 underwent pulsed RF (180sec, with a fixed temperature at 42C, twice) on the suprascapular nerve, and the other group, 2, underwent nerve block with bupivacaine (5ml). After the procedure, patients were evaluated for 3 months regarding pain intensity, shoulder range of motion and dose of rescue opioids.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years old
* Chronic shoulder pain (more than 3 months)
* Clinical and imaging diagnosis: rotator cuff injury, adhesive capsulitis, supraspinatus, tendinopathy, bicipital tendinitis, impingement syndrome, subscapularis tendinopathy, , subacromial and subdeltoid arthrosis, acromioclavicular arthrosis, subdeltoid subacromial bursitis
* Pain intensity ≥4 on movement, on a numerical scale from zero to 10 (where zero means no pain and 10 the most intense pain imaginable).

Exclusion Criteria:

* Arrhythmia
* Cognitive change (inability to answer questions)
* Psychiatric illness
* Infection at the site of the procedure
* Coagulopathy,
* Use of anticoagulants
* Hypersensitivity to medications
* Pregnant
* Use of pacemaker

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Comparison of pain intensity after application of pulsed RF in the suprascapular nerve versus injection of a local anesthetic. | 12 months
  Comparison of pain intensity after application of pulsed RF to the suprascapular nerve and after injection of a local anesthetic. The numerical pain scale (Visual Analogue Scale - VAS) at rest and during movement was used. This scale (VAS) ranges from 1 to 10, with 1 representing mild pain and 10 representing severe pain.

SECONDARY OUTCOMES:
To assess the range of motion of the shoulder joint | 12 months
  To assess the range of motion of the shoulder joint. A goniometer was used to assess the range of motion.
Need for additional analgesic. | 12 months
  Assessment of the need for additional analgesics according to pain. Pain was measured using the Visual Analogue Scale, ranging from 1 to 10, with 1 representing mild pain and 10 representing severe pain.
Duration of the analgesic effect. | 12 months
  Pain was assessed using the numerical pain scale (Visual Analogue Scale - VAS). The participant was asked to respond on a scale of 1 to 10, with 1 representing mild pain and 10 representing severe pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of Sao Paulo - Hospital Sao Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No